CLINICAL TRIAL: NCT01409109
Title: Database Registry to Examine Brain Connections and Brain Function in Mental Disorders and Neural Network Biomarkers for Relational Memory and Psychosis in Schizophrenia
Brief Title: Database Registry for Neural Network Biomarkers in Psychosis
Acronym: Imaging
Status: Active, not recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Carol A. Tamminga, Principal Investigator, University of Texas Southwestern Medical Center
Other Study IDs: STU 062010-095; 1R01MH083957-01A2 (NIH); 1K23MH102656-01A1 (NIH)
Record Dates: First submitted 2011-06-29; First posted 2011-08-03 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective; Neuroimaging; Magnetic Resonance Imaging (MRI); Functional Magnetic Resonance Imaging (fMRI); Spectroscopy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (2):
- Patient volunteers: This group is comprised of persons with Schizophrenia and Schizoaffective.
- Healthy volunteers: This group is comprised of individuals who have no current or past psychiatric diagnosis.

SUMMARY:
Several observations have been made with magnetic resonance imaging (MRI) that characterize brain connections and brain function in individuals with schizophrenia and other mental disorders. For example, research investigating schizophrenia focuses on the dysfunction of connections within and between the medial temporal lobe and the prefrontal cortex as well as other pertinent brain regions. This database registry will allow for the collection of clinical interview data, behavioral data, blood, magnetic resonance imaging (MRI) data, and functional magnetic resonance imaging (fMRI) data on individuals with and without mental disorders to better understand how connections in the brain and various brain regions function differently while volunteers perform various cognitive tasks. This is an observational study that is being conducted to collect data and place it in a registry for current and future investigational questions related to imaging in mental disorders.

DETAILED DESCRIPTION:
The proposed project entails the collection of clinical interview data, behavioral data, blood, magnetic resonance imaging (MRI) data, and functional magnetic resonance imaging (fMRI) data from 1000 volunteers, both patient volunteers and healthy normal volunteers. These data will be used for current and future investigations to better understand how the brains of those with mental disorders process differently that brains of healthy volunteers. The volunteers will undergo a series of clinical interviews to determine their diagnosis, behavioral task training, medical workup, and standard structural and functional magnetic resonance imaging. No changes will be made to the patient volunteers' medications or treatment regimes as part of the study. Data will be collected for all volunteer groups based on their performance on a variety of computer-mediated cognitive tasks. The volunteers will be trained to criteria on the tasks, at which point they will have the option to complete the MRI and fMRI portions of the study. Standard and functional MR images of the entire brain will be acquired while volunteers perform cognitive tasks thought to activate the medial temporal lobe and other pertinent brain regions. While participating in the task portion of the fMRI, visual stimulation (images) will be presented via back-projection from a high-resolution video projector (Epson 7000 series) with adjustable zoom. Volunteers will be asked to push a button on a handheld button box to record their responses as learned during training. For the non-task, resting portions of the fMRI, volunteers will be asked to stay relaxed and alert. In conjunction with one of the fMRI scans we will also conduct a cerebral blood volume (CBV) MRI to investigate blood perfusion in the medial temporal lobe of volunteers with mental illness to compare to normal control volunteers.

The proposed project will evaluate brain connectivity during cognitive tasks, including novelty detection, encoding and retrieval of associations between individual stimuli, and during other cognitive tasks thought to produce abnormal fMRI activations in volunteers with mental disorders. One example of a cognitive task is conducted as follows. Volunteers are shown a series of one-syllable nouns and asked to internally associate a second noun to the presented word (e.g. "station" to the presented word "train"). They press a response button when they have made a successful word association. Subsequently, volunteers are presented with a mixture of the previously encoded words and a new set of one-syllable nouns. Volunteers press one response button for previously presented words and another button for novel (new) words. fMRI scans for both parts of this task are acquired in the time between stimulus presentation and the press of the button. In another example of a cognitive task, volunteers are shown a novel series of faces paired with names and are instructed to remember the name for each face. In a subsequent period, volunteers attempt to remember which name goes to which face. The fMRI scans are acquired during both encoding and retrieval of the face-name pairs. These two described tasks are representative of the tasks to be used in terms of their difficulty and the effort required of the volunteers. In addition, "resting" and "control" tasks will be used to establish a baseline of brain activity against which we may then compare activity during our task of interest. Volunteers will receive instructions on task performance and will practice tasks prior to scanning in order to eliminate the novelty of the task itself as a potential confound. While the appointment time for a scan may take several hours, the volunteer will be in the scanner between 60 and 120 minutes depending on the specific memory task that is being administered at that visit. Any volunteer may receive training and be scanned on more than one task, but no volunteer will be kept in the scanner for longer than 120 minutes in any given session. Volunteers may also be asked to undergo one or two 60-minute MR Spectroscopy scans conducted on the 3Tesla (3T) or 7Tesla (7T) scanner. In this scan we will measure the levels of different brain compounds, such as neurotransmitters (e.g. glutamate, gamma aminobutyric acid [GABA]) or endogenous brain metabolites (e.g., N-acetyl -aspartate)in various brain regions, to non-invasively study tissue biochemistry.

ELIGIBILITY:
Inclusion Criteria:

Volunteers with Schizophrenia or other mental illness

* Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) diagnosis of Schizophrenia or Schizoaffective disorder
* Competent to give informed consent
* All races and ethnicities
* Eyesight corrected to 20-40 or better
* Able to read, speak, and understand English

Healthy volunteers

* No past or current severe mental illness
* All races and ethnicities
* Eyesight corrected to 20-40 or better
* Able to read, speak, and understand English

Exclusion Criteria:

Volunteers with schizophrenia or other mental illness

* Diagnosis of an organic brain disease
* Diagnosis of DSM-IV-TR alcohol or substance abuse within the last month or DSM-IV-TR alcohol or substance dependence within the last three months
* Serious, unstable medical illness
* History of serious head injury
* Pregnant women

Healthy volunteers

* History of psychiatric illness
* Current use of psychoactive drugs excluding nicotine and caffeine
* Diagnosis of an organic brain disease
* Serious, unstable medical illness
* History of serious head injury
* Pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals who have been diagnosed with the following disorders will be enrolled in this study: Schizophrenia and Schizoaffective disorder.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-03; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Differences in hippocampal subfield activation between people with schizophrenia (or schizoaffective disorder) and healthy volunteers | Participants will be assessed over the course of 4-6 weeks, until all study procedures are complete
  This study will investigate the alterations in the medial temporal lobe, specifically the differences in hippocampal subfield activation, between patients with psychosis (Schizophrenia and Schizoaffective disorder), their relatives and normal volunteers. We hypothesize that there will be an increase in perfusion and a decrease in subfield activation in the people with psychosis.

SECONDARY OUTCOMES:
Differences in glutamate neurotransmitters and glutamatergic function between people with schizophrenia (or schizoaffective disorder) and with healthy volunteers | Participants will be assessed over the course of 4-6 weeks, until all study procedures are complete
  We aim to measure glutamate-related neurochemical profiles in schizophrenia using proton magnetic resonance spectroscopy (MRS) 7T. We will measure several brain metabolites, including glutamate, glutamine, GABA, glycine, N-acetylaspartyl-glutamate, glutathione, and myo-inositol, in addition to other major signals in brain MRS (i.e., N-acetylaspartate, creatine and choline), in anterior cingulate cortex (ACC) and dorsolateral prefrontal cortex (DLPFC) in volunteers with schizophrenia (SZ) and normal volunteers (NV).

CONTACTS AND LOCATIONS:
Overall Officials: Carol A. Tamminga, M.D., Principal Investigator — UT Southwestern; Elena Ivleva, M.D., Ph.D., Principal Investigator — UT Southwestern
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- See also: Division of Translational Neuroscience Research in Schizophrenia — http://www.utsouthwestern.edu/labs/schizophrenia/